CLINICAL TRIAL: NCT05584306
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase Ib Study to Determine the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of Recombinant Anti-IL-5 Humanized Monoclonal Antibody Therapy in Adult Subjects With Severe Eosinophilic Asthma
Brief Title: A Dose Ranging Placebo-controlled Double-blind Study to Evaluate the Safety, Pharmacokinetics and Efficacy of 610 in Participants With Severe Eosinophilic Asthma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SSGJ-610-BA-I/II-01
Record Dates: First submitted 2022-10-09; First posted 2022-10-18 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Asthma
Keywords: Asthma; Eosinophilic asthma; Exacerbations; 610; Placebo
MeSH Terms: conditions — Asthma; Pulmonary Eosinophilia | interventions — Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 610 30mg group (Experimental): 610 30 mg administered subcutaneously every 4 weeks
  Interventions: Drug: 610 30mg group
- 610 100mg group (Experimental): 610 100 mg administered subcutaneously every 4 weeks
  Interventions: Drug: 610 100mg group
- 610 300mg group (Experimental): 610 300mg administered subcutaneously every 4 weeks
  Interventions: Drug: 610 300mg group
- Placebo 30mg group (Placebo Comparator): placebo subcutaneous (SC) Q4W，8 times
  Interventions: Other: Placebo 30mg group
- Placebo 100mg group (Placebo Comparator): placebo subcutaneous (SC) Q4W，8 times
  Interventions: Other: Placebo 100mg group
- Placebo 300mg group (Placebo Comparator): placebo subcutaneous (SC) Q4W，8 times
  Interventions: Other: Placebo 300mg group

INTERVENTIONS:
Drug: 610 30mg group — 610 30mg subcutaneous (SC) Q4W，8 times
  Arms: 610 30mg group
Drug: 610 100mg group — 610 100mg subcutaneous (SC) Q4W，8 times
  Arms: 610 100mg group
Drug: 610 300mg group — 610 300mg subcutaneous (SC) Q4W，8 times
  Arms: 610 300mg group
Other: Placebo 30mg group — placebo subcutaneous (SC) Q4W，8 times
  Arms: Placebo 30mg group
Other: Placebo 100mg group — placebo subcutaneous (SC) Q4W，8 times
  Arms: Placebo 100mg group
Other: Placebo 300mg group — placebo subcutaneous (SC) Q4W，8 times
  Arms: Placebo 300mg group

SUMMARY:
This study will assess the safety, tolerability, pharmacokinetics and preliminary efficacy of 610 as an adjunctive therapy in adult subjects with severe eosinophilic asthma.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled study to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of 610 in adults with severe eosinophilic asthma. Plan to recruit 24 subjects, and the subjects divided into 3 groups: 610 30mg group，100mg group, 610 300mg group，8 subjects in each dose group, of which 6 received the trial drug and 2 received placebo. The study is divided into screening period of 2 weeks, treatment period of 32 weeks and follow-up period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with asthma for ≥12 months
* Within 3 months before screening, treatment with medium to high dose inhaled corticosteroid（ICS，inhaled fluticasone at a dosage of at least 500 μg, or equivalent, daily.）and at least one other additional controller medication, such as long-acting β₂ receptor agonist (LABA), leukotriene receptor antagonist (LTRA), theophylline, long-acting Anticholinergic drugs (LAMA), etc. Those medicine must be stable for ≥ 28 days prior to screening and baseline and must continue without dosage changes throughout the study
* In the past 12 months prior to screening， at least one time asthma exacerbations history
* Pre-bronchodilator FEV1 <80% predicted value
* Asthma-related blood eosinophils ≥ 150 cells/μL within 3 months before administration

Exclusion Criteria:

* With clinically important lung diseases other than asthma that may affect safety or efficacy and evaluated by investigator. This includes lung infection, chronic obstructive pulmonary disease, bronchiectasis, hypersensitivity pneumonitis, pulmonary fibrosis, Allergic bronchopulmonary aspergillosis, etc.
* With other conditions that could lead to elevated eosinophils such as hypereosinophilic syndromes, eosinophilic granulomatosis with polyangiitis (EGPA), or eosinophilic esophagitis
* In past 12 months prior to screening，patients has done bronchial thermoplasty or radiotherapy or plan to do it during of the trial
* with severe cardiac disease or uncontrolled or severe cardiac arrhythmia
* poorly controlled systemic disease
* Active infection 7 day before screening
* Parasitic infection within 6 months before screening
* At screening, HBsAg or HCV Ab or HIV Ab or TP Ab positive; HBsAg or HCV Ab positive need to be further tested of HBV DNA titer detection or HCV RNA detection (More than normal value range needs to be excluded)
* Subjects who have received any monoclonal antibody treatment of anti IL-4Ror anti-IL-5/5R
* Vaccination history with live vaccines (including live attenuated vaccines) within 4 weeks before screening, or plan to receive during of the trial
* Participated in any interventional clinical trial and received intervention within 3 months before screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-12-06 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Adverse events(AEs) | From Day 0 to Day 308
  The incidence and severity of AEs, including SAEs, as well as clinical symptoms, and any abnormalities of vital signs, physical examinations#electrocardiogram#laboratory tests and, etc.

SECONDARY OUTCOMES:
Pharmacokinetics-Tmax | From Day 0 to Day 308
  Time to Cmax of 610
Pharmacokinetics-AUC0-last | From Day 0 to Day 308
  Area under the concentration-time curve from time 0 to last time point after 610 subcutaneous
Pharmacokinetics-AUC0-inf | From Day 0 to Day 308
  Area under the concentration-time curve from time 0 to infinity after 610 subcutaneous
Pharmacokinetics-Cmax | From Day 0 to Day 308
  Maximum observed concentration of 610
Pharmacokinetics-CL/F | From Day 0 to Day 308
  Apparent clearance of 610
Pharmacokinetics-Vz/F | From Day 0 to Day 308
  Apparent volume of distribution during terminal phase of 610
Pharmacokinetics-t1/2 | From Day 0 to Day 308
  Terminal elimination half-life of 610
Pharmacodynamics-Eosinophils | From Day 0 to Day 308
  Absolute eosinophils account and change from baseline in percentage
Anti-drug-antibody | From Day 0 to Day 308
  The percentage of subjects with positive ADA titers over time for 610
Number of asthma exacerbation | From Day 0 to Day 308
  Asthma exacerbation are defined as worsening of asthma which required use of systemic corticosteroids (≥3 days. For maintenance of systemic corticosteroids, at least double the existing maintenance dose for at least 3 days was required) and/or hospitalization and/or emergency department (ED) visits.
Changes from baseline in pre-bronchodilator forced expiratory volume in one second (FEV1) | From Day 0 to Day 308
  FEV1 is defined as the volume of air expelled from the lungs in 1 second. Pre-bronchodilator FEV1 measurements were taken by spirometry.
Percentage change from baseline in pre-bronchodilator forced expiratory volume in one second (FEV1) | From Day 0 to Day 308
  Percentage of FEV1 will be measured using spirometry.
Time to first asthma exacerbation event | From Day 0 to Day 308
  Asthma exacerbation are defined as worsening of asthma which required use of systemic corticosteroids (≥3 days. For maintenance of systemic corticosteroids, at least double the existing maintenance dose for at least 3 days was required) and/or hospitalization and/or emergency department (ED) visits.
Number of asthma exacerbations requiring hospitalization (including intubation and ICU admission) or emergency room visits (not conversion to hospitalization) | From Day 0 to Day 308
  Asthma exacerbations that are associated with a hospitalization or an emergency room visit.
Number of asthma exacerbations requiring hospitalization (including intubation and ICU admission) | From Day 0 to Day 308
  Asthma exacerbations that are associated with a hospitalization.
Change from baseline in Asthma Control Questionnaire score | From Day 0 to Day 308
  The ACQ has 7 questions- the first 5 items assess the most common asthma symptoms plus 6. short-acting bronchodilator use and 7. FEV1 (pre-bronchodilator use, % and % predicted use). Patients are asked to recall how their asthma has been during the previous week and to respond to the symptom questions on a 7-point scale (0=no impairment, 6= maximum impairment).
Change From Baseline in the St. George's Respiratory Questionnaire Total Score | From Day 0 to Day 308
  The St. George's Respiratory Questionnaire is an established instrument, comprising 50 questions, evaluating symptoms, activity, and impacts; to measure Quality of Life in participants with diseases of airway obstruction and to elicit the participant's opinion of his/her health.

CONTACTS AND LOCATIONS:
Overall Officials: Qinghong Zhou, MD, Study Director — Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd.; Xin Zhou, MD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine; Min Zhang, MD, Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No